CLINICAL TRIAL: NCT02571660
Title: Efficacy of Vitamin D on the Clinical Management of Pediatric Patients With Asthma in the Hospital General Naval de Alta Especialidad
Brief Title: Efficacy of Vitamin D on the Clinical Management of Pediatric Patients With Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government)
Responsible Party: Principal Investigator, Dr. Jorge Ivan Valencia Moncada, Dr. Emmanuelle Dexeus Gabriel Fernandez Vera, Hospital General Naval de Alta Especialidad - Escuela Medico Naval
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGNAE 05
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Asthma
Keywords: vitamin d levels; exacerbation of asthma; asthma control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional treatment (Active Comparator): GINA treatment fot asthma +vit.D low supplementation dose
  Interventions: Drug: GINA treatment fot asthma +vit.D low supplementation dose
- conventional treatment + vitamin D3 (Experimental): GINA treatment fot asthma +vit.D high supplementation dose
  Interventions: Drug: GINA treatment fot asthma +vit.D high supplementation dose

INTERVENTIONS:
Drug: GINA treatment fot asthma +vit.D low supplementation dose — Dose of 400 IU of vitamin D3 every 24 hours for 1 year + the standard treatment for asthma,
  Other Names: SD group
  Arms: conventional treatment
Drug: GINA treatment fot asthma +vit.D high supplementation dose — Dose of 1600 IU of vitamin D3 be allocated each 24 hours for 1 year + standard treatment for asthma
  Other Names: TD group
  Arms: conventional treatment + vitamin D3

SUMMARY:
Asthma is a disease that represents a public health problem worldwide, there are several barriers, especially in pediatric patients with this disease, them, prevent the adequate control of their condition, in addition every day there are new processing aids for this entity; within these novel research we founded the relationship between decreased vitamin D serum levels and his role in the regulating of the immune response, also this relationship in the pathophysiology of this disease and responses in the event of infectious diseases of the respiratory tract which can exacerbate symptoms in pediatric patients. We have been some of clinical trials with the aim of improving serum levels of vitamin D in asthmatic patients, however, these studies have different sources of bias and thus far there is no solid evidence that favors or denies the relationship between asthma and vitamin D, this paper aims to help generate this evidence to improve clinical management of these patients and their lung function and increase the free time crisis.

In this trial two study groups which are divided for each of the interventions described below:

Group low supplementation dose: 1 tablet of 400 IU was administered every 24 hours via oral, regardless of time or if it is before or after food, preferably in the morning to improve adherence to treatment, will be completed one year of treatment without suspension.

Group high supplementation dose: 1 tablet of 1600 IU should be administered every 24 hours via oral, regardless of time or if it is before or after food, preferably in the morning to improve adherence to treatment, will be completed one year of treatment without suspension thereof.

DETAILED DESCRIPTION:
There are several potential mechanisms that have been described both in vitro models and in vivo models in which has been linked to asthma control with elevated levels of vitamin D in serum. These mechanisms include structural effects in the lungs, immunomodulation, modulation of smooth muscle response to level and effect on bronchial response to inhaled medicines to treat asthma.

* Structural mechanisms Studies were conducted in rats of 50 days old, lung compliance was measured and decreased it in rats whose mothers had a diet of deprivation of vitamin D compared to those rats whose mothers received vitamin supplementation was observed. In human groups, pulmonary function tests at age 6 were carried out, and there was a significant difference between children with mothers with vitamin D deficiency during pregnancy and children whose mothers had normal levels during pregnancy. These findings suggest that there is a strong relationship between lung embryonic development serum level of vitamin D and therefore this plays a key role in the structural development of the airways
* Anti-inflammatory Mechanisms Within these mechanisms, they are significantly inhibiting pro-inflammatory cytokines such as interleukin-6 and tumor necrosis factor alpha (TNF-A) by way of inhibition of MAP 38 produced by monocytes. Another such mechanism is the inhibition of transcription factor (necrosis factor kappa-beta). We observed a decrease in the phosphorylation and production of reactive oxygen species with the addition of 1-25 dihydroxyvitamin D levels which leads to less inflammatory damage in the respiratory epithelium.
* Immunomodulation Effects occur in both innate immunity and adaptive, innate immunity in the effect of 1,25 hydroxyvitamin D has an effect on the reduction of inflammatory cytokines and in the decreased expression of Toll-like receptors monocytes. Also active antimicrobial peptides such as defensin 2 and 4 and the human defensin cathecidina 18, studies where low levels of vitamin D are associated and low levels of this peptide
* Effects on helper T lymphocytes Molecular effects, vitamin D levels are associated with decreased circulating IgE as well as decreasing the TH1 response and therefore TH2, however the role of vitamin D on these cells is unclear, and some studies have shown the prevalence of TH2 response in patients with adequate levels of Vitamin D, however the decrease in the inflammatory response and the production of cytokines such as IL 12 has shown that vitamin D it modulates the response that causes pathogenesis Asthma
* Decrease in early infections or severity The previously mentioned effects on adaptive and innate immunity may decrease the risk of early respiratory tract infections, which have been associated in the first years of life with a high incidence of wheezing. In Hawaiian children under age 5 suffering from rickets incidence of respiratory tract diseases and wheezing it was higher than that of the population without vitamin D deficiency

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 7 to 15 years regardless of sex diagnosed with asthma by clinical suspicion and accurate diagnosis by spirometry positive flow limitation with bronchodilator reversibility
* Controlled pediatric Pneumology service Patients
* Patients whose parents accept the child's participation by signing the informed consent. For children over 12 years the least sign the informed consent personally

Exclusion Criteria:

* Patients with hypocalcemia or hypercalcemia
* Patients with kidney diseases such as kidney stones, hypercalciuria, renal tubular acidosis
* Patients with moderate to severe malnutrition

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Free lapse of asthma exacerbation | 1 year
  Compare between the group treated with vitamin D at doses of 4 RDA combined with standard treatment of asthma versus the group treated with vitamin D at doses of 1 RDA combined with standard treatment group:
  •Free lapse of asthma exacerbation in asthmatic patients 7-15 years of age

SECONDARY OUTCOMES:
Clinical control of asthma | 1 year
  Compare between the groups the clinical control of asthma with the questionary: asthma control test
Lung function | 1 year
  Compare both groups improved lung function measured by spirometry using as parameter FEV 1
Vitamin D serum levels | 1 year
  Determine serum levels of vitamin D , basal and after treatment in patients included in this study
Season levels of vitamin D | 1 year
  Compare serum levels of vitamin D in different seasons
Serum vitamin D levels and clinical control of asthma | 1 year
  to determine the correlation between serum levels of vitamin d with clinical asthma control

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Dexeus Gabriel Fernandez, pediatrician, Principal Investigator — Hospital General Naval de Alta Especialidad - Escuela Medico Naval
Locations (1):
- Hospital General Naval de Alta Especialidad, Distrito Federal, Mexico City, Mexico

REFERENCES:
- [Background] Papadopoulos NG, Arakawa H, Carlsen KH, Custovic A, Gern J, Lemanske R, Le Souef P, Makela M, Roberts G, Wong G, Zar H, Akdis CA, Bacharier LB, Baraldi E, van Bever HP, de Blic J, Boner A, Burks W, Casale TB, Castro-Rodriguez JA, Chen YZ, El-Gamal YM, Everard ML, Frischer T, Geller M, Gereda J, Goh DY, Guilbert TW, Hedlin G, Heymann PW, Hong SJ, Hossny EM, Huang JL, Jackson DJ, de Jongste JC, Kalayci O, Ait-Khaled N, Kling S, Kuna P, Lau S, Ledford DK, Lee SI, Liu AH, Lockey RF, Lodrup-Carlsen K, Lotvall J, Morikawa A, Nieto A, Paramesh H, Pawankar R, Pohunek P, Pongracic J, Price D, Robertson C, Rosario N, Rossenwasser LJ, Sly PD, Stein R, Stick S, Szefler S, Taussig LM, Valovirta E, Vichyanond P, Wallace D, Weinberg E, Wennergren G, Wildhaber J, Zeiger RS. International consensus on (ICON) pediatric asthma. Allergy. 2012 Aug;67(8):976-97. doi: 10.1111/j.1398-9995.2012.02865.x. Epub 2012 Jun 15. PMID 22702533
- [Result] Hill VL, Wood PR. Asthma epidemiology, pathophysiology, and initial evaluation. Pediatr Rev. 2009 Sep;30(9):331-5; quiz 335-6. doi: 10.1542/pir.30-9-331. PMID 19726699
- [Result] Wood PR, Hill VL. Practical management of asthma. Pediatr Rev. 2009 Oct;30(10):375-85; quiz 385. doi: 10.1542/pir.30-10-375. PMID 19797480
- [Result] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Result] Worldwide variations in the prevalence of asthma symptoms: the International Study of Asthma and Allergies in Childhood (ISAAC). Eur Respir J. 1998 Aug;12(2):315-35. doi: 10.1183/09031936.98.12020315. PMID 9727780
- [Result] Murphy DM, O'Byrne PM. Recent advances in the pathophysiology of asthma. Chest. 2010 Jun;137(6):1417-26. doi: 10.1378/chest.09-1895. PMID 20525652
- [Result] Berry M, Morgan A, Shaw DE, Parker D, Green R, Brightling C, Bradding P, Wardlaw AJ, Pavord ID. Pathological features and inhaled corticosteroid response of eosinophilic and non-eosinophilic asthma. Thorax. 2007 Dec;62(12):1043-9. doi: 10.1136/thx.2006.073429. Epub 2007 Mar 13. PMID 17356056
- [Result] Majak P, Olszowiec-Chlebna M, Smejda K, Stelmach I. Vitamin D supplementation in children may prevent asthma exacerbation triggered by acute respiratory infection. J Allergy Clin Immunol. 2011 May;127(5):1294-6. doi: 10.1016/j.jaci.2010.12.016. Epub 2011 Feb 18. No abstract available. PMID 21315433
- [Result] Bar Yoseph R, Livnat G, Schnapp Z, Hakim F, Dabbah H, Goldbart A, Bentur L. The effect of vitamin D on airway reactivity and inflammation in asthmatic children: A double-blind placebo-controlled trial. Pediatr Pulmonol. 2015 Aug;50(8):747-53. doi: 10.1002/ppul.23076. Epub 2014 Jul 2. PMID 24989842
- [Result] Castro M, King TS, Kunselman SJ, Cabana MD, Denlinger L, Holguin F, Kazani SD, Moore WC, Moy J, Sorkness CA, Avila P, Bacharier LB, Bleecker E, Boushey HA, Chmiel J, Fitzpatrick AM, Gentile D, Hundal M, Israel E, Kraft M, Krishnan JA, LaForce C, Lazarus SC, Lemanske R, Lugogo N, Martin RJ, Mauger DT, Naureckas E, Peters SP, Phipatanakul W, Que LG, Sheshadri A, Smith L, Solway J, Sullivan-Vedder L, Sumino K, Wechsler ME, Wenzel S, White SR, Sutherland ER; National Heart, Lung, and Blood Institute's AsthmaNet. Effect of vitamin D3 on asthma treatment failures in adults with symptomatic asthma and lower vitamin D levels: the VIDA randomized clinical trial. JAMA. 2014 May;311(20):2083-91. doi: 10.1001/jama.2014.5052. PMID 24838406
- [Result] Martineau AR, MacLaughlin BD, Hooper RL, Barnes NC, Jolliffe DA, Greiller CL, Kilpin K, McLaughlin D, Fletcher G, Mein CA, Hoti M, Walton R, Grigg J, Timms PM, Rajakulasingam RK, Bhowmik A, Rowe M, Venton TR, Choudhury AB, Simcock DE, Sadique Z, Monteiro WR, Corrigan CJ, Hawrylowicz CM, Griffiths CJ. Double-blind randomised placebo-controlled trial of bolus-dose vitamin D3 supplementation in adults with asthma (ViDiAs). Thorax. 2015 May;70(5):451-7. doi: 10.1136/thoraxjnl-2014-206449. Epub 2015 Feb 27. PMID 25724847
- [Result] Unuvar T, Buyukgebiz A. Nutritional rickets and vitamin D deficiency in infants, children and adolescents. Pediatr Endocrinol Rev. 2010 Mar-Apr;7(3):283-91. PMID 20526242
- [Result] Brehm JM, Schuemann B, Fuhlbrigge AL, Hollis BW, Strunk RC, Zeiger RS, Weiss ST, Litonjua AA; Childhood Asthma Management Program Research Group. Serum vitamin D levels and severe asthma exacerbations in the Childhood Asthma Management Program study. J Allergy Clin Immunol. 2010 Jul;126(1):52-8.e5. doi: 10.1016/j.jaci.2010.03.043. Epub 2010 Jun 9. PMID 20538327
- [Result] Dabbah H, Bar Yoseph R, Livnat G, Hakim F, Bentur L. Bronchial Reactivity, Inflammatory and Allergic Parameters, and Vitamin D Levels in Children With Asthma. Respir Care. 2015 Aug;60(8):1157-63. doi: 10.4187/respcare.03763. Epub 2015 Apr 21. PMID 25899478
- [Result] Bener A, Ehlayel MS, Tulic MK, Hamid Q. Vitamin D deficiency as a strong predictor of asthma in children. Int Arch Allergy Immunol. 2012;157(2):168-75. doi: 10.1159/000323941. Epub 2011 Oct 6. PMID 21986034
- [Result] Alshahrani F, Aljohani N. Vitamin D: deficiency, sufficiency and toxicity. Nutrients. 2013 Sep 13;5(9):3605-16. doi: 10.3390/nu5093605. PMID 24067388
- [Result] Ginde AA, Sutherland ER. Vitamin D in asthma: panacea or true promise? J Allergy Clin Immunol. 2010 Jul;126(1):59-60. doi: 10.1016/j.jaci.2010.05.030. No abstract available. PMID 20620566
- [Result] Gergen PJ, Teach SJ, Mitchell HE, Freishtat RF, Calatroni A, Matsui E, Kattan M, Bloomberg GR, Liu AH, Kercsmar C, O'Connor G, Pongracic J, Rivera-Sanchez Y, Morgan WJ, Sorkness CA, Binkley N, Busse W. Lack of a relation between serum 25-hydroxyvitamin D concentrations and asthma in adolescents. Am J Clin Nutr. 2013 Jun;97(6):1228-34. doi: 10.3945/ajcn.112.046961. Epub 2013 Apr 17. PMID 23595876
- [Result] Goleva E, Searing DA, Jackson LP, Richers BN, Leung DY. Steroid requirements and immune associations with vitamin D are stronger in children than adults with asthma. J Allergy Clin Immunol. 2012 May;129(5):1243-51. doi: 10.1016/j.jaci.2012.01.044. Epub 2012 Feb 11. PMID 22330698
- [Result] Poon AH, Mahboub B, Hamid Q. Vitamin D deficiency and severe asthma. Pharmacol Ther. 2013 Nov;140(2):148-55. doi: 10.1016/j.pharmthera.2013.06.006. Epub 2013 Jun 18. PMID 23792089
- [Result] Chinellato I, Piazza M, Sandri M, Peroni D, Piacentini G, Boner AL. Vitamin D serum levels and markers of asthma control in Italian children. J Pediatr. 2011 Mar;158(3):437-41. doi: 10.1016/j.jpeds.2010.08.043. Epub 2010 Sep 26. PMID 20870246
- [Result] Hatami G, Ghasemi K, Motamed N, Firoozbakht S, Movahed A, Farrokhi S. Relationship between Vitamin D and Childhood Asthma: A Case-Control Study. Iran J Pediatr. 2014 Dec;24(6):710-4. Epub 2014 Nov 7. PMID 26019776
- [Result] Dogru M, Kirmizibekmez H, Yesiltepe Mutlu RG, Aktas A, Ozturkmen S. Clinical effects of vitamin D in children with asthma. Int Arch Allergy Immunol. 2014;164(4):319-25. doi: 10.1159/000366279. Epub 2014 Sep 23. PMID 25277142
- [Result] Maguire JL, Birken CS, Loeb MB, Mamdani M, Thorpe K, Hoch JS, Mazzulli T, Borkhoff CM, Macarthur C, Parkin PC; TARGet Kids! Collaboration. DO IT Trial: vitamin D Outcomes and Interventions in Toddlers - a TARGet Kids! randomized controlled trial. BMC Pediatr. 2014 Feb 8;14:37. doi: 10.1186/1471-2431-14-37. PMID 24506910
- [Result] Majak P, Rychlik B, Stelmach I. The effect of oral steroids with and without vitamin D3 on early efficacy of immunotherapy in asthmatic children. Clin Exp Allergy. 2009 Dec;39(12):1830-41. doi: 10.1111/j.1365-2222.2009.03357.x. Epub 2009 Oct 7. PMID 19817753
- [Result] Beigelman A, Zeiger RS, Mauger D, Strunk RC, Jackson DJ, Martinez FD, Morgan WJ, Covar R, Szefler SJ, Taussig LM, Bacharier LB; Childhood Asthma Research and Education (CARE) Network of the National Heart, Lung, and Blood Institute. The association between vitamin D status and the rate of exacerbations requiring oral corticosteroids in preschool children with recurrent wheezing. J Allergy Clin Immunol. 2014 May;133(5):1489-92, 1492.e1-3. doi: 10.1016/j.jaci.2014.02.024. Epub 2014 Apr 1. No abstract available. PMID 24698320
- [Result] Leung TF, Wang SS, Tang MF, Kong AP, Sy HY, Hon KL, Chan JC, Wong GW. Childhood asthma and spirometric indices are associated with polymorphic markers of two vitamin D 25-hydroxylase genes. Pediatr Allergy Immunol. 2015 Jun;26(4):375-82. doi: 10.1111/pai.12392. PMID 25845986
- [Result] Fares MM, Alkhaled LH, Mroueh SM, Akl EA. Vitamin D supplementation in children with asthma: a systematic review and meta-analysis. BMC Res Notes. 2015 Feb 3;8:23. doi: 10.1186/s13104-014-0961-3. PMID 25643669
- [Result] Cassim R, Russell MA, Lodge CJ, Lowe AJ, Koplin JJ, Dharmage SC. The role of circulating 25 hydroxyvitamin D in asthma: a systematic review. Allergy. 2015 Apr;70(4):339-54. doi: 10.1111/all.12583. PMID 25631639
- [Result] Garcia de Tena J, El Hachem Debek A, Hernandez Gutierrez C, Izquierdo Alonso JL. The role of vitamin D in chronic obstructive pulmonary disease, asthma and other respiratory diseases. Arch Bronconeumol. 2014 May;50(5):179-84. doi: 10.1016/j.arbres.2013.11.023. Epub 2014 Jan 18. English, Spanish. PMID 24447429
- [Result] Luong Kv, Nguyen LT. The role of vitamin D in asthma. Pulm Pharmacol Ther. 2012 Apr;25(2):137-43. doi: 10.1016/j.pupt.2012.02.003. PMID 22532985
- [Result] Kerley CP, Elnazir B, Faul J, Cormican L. Vitamin D as an adjunctive therapy in asthma. Part 1: A review of potential mechanisms. Pulm Pharmacol Ther. 2015 Jun;32:60-74. doi: 10.1016/j.pupt.2015.02.004. Epub 2015 Feb 28. PMID 25732539
- [Result] Kerley CP, Elnazir B, Faul J, Cormican L. Vitamin D as an adjunctive therapy in asthma. Part 2: A review of human studies. Pulm Pharmacol Ther. 2015 Jun;32:75-92. doi: 10.1016/j.pupt.2015.02.010. Epub 2015 Mar 5. PMID 25749414